CLINICAL TRIAL: NCT01224444
Title: Complete Histologic Resection of Adenomatous Polyps? (Complete Adenoma REsection Trial - CARE Trial)
Brief Title: Complete Histologic Resection of Adenomatous Polyps?
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Heiko Pohl, Principal Investigator, White River Junction Veterans Affairs Medical Center
Other Study IDs: DMS-21237
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-12

CONDITIONS: Adenomatous Polyps
Keywords: colon polyps; adenoma resection; colon cancer screening; colonoscopy
MeSH Terms: conditions — Adenomatous Polyps; Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies will be taken from resection margins: 2 biopsies will be obtained from opposite margins for polyps 5-9mm, and 4 biopsies will be taken for polyps 10-20mm from all four quadrants of the resection margins.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All adenomatous polyps: Standard polypectomy snare of adenomatous polyps (included serrated adenomas) from ≤5mm to ≤20mm.
  Interventions: Other: standard polypectomy snare

INTERVENTIONS:
Other: standard polypectomy snare — Electrocautery snare resection of sessile colonic polyps

SUMMARY:
Colorectal cancer is the second most common cause of cancer death in the US. Colonoscopy is considered the best test colorectal cancer screening. It allows resection of adenomatous polyps (a known cancer precursor) and thus, interrupt the adenoma-carcinoma sequence. Despite the potential benefit of screening colonoscopy recent studies have reported cases of colorectal cancers in a short interval after prior screening or surveillance colonoscopies. One possible cause of such interval cancers may be incomplete resection of adenomatous polyps and hence ongoing growth and cancer development in such lesions. Complete resection may be particularly important for polyps of at least 5mm in size as up 10% of such polyps higher risk lesions as villous adenoma, tubulovillous adenoma, high grade dysplasia, or early carcinoma.

Although adenoma resection of sessile and flat adenomatous polyps between 5 and 20mm is believed to be well standardized data on complete resection of adenomatous tissue are sparse. This may be related to the assumption that using a snare with electro-cautery will successfully remove the polyp and cauterize remaining marginal adenomatous tissue and hence completely remove and or destroy the lesion.

The investigators are interested in examining how often sessile adenomatous polyps between 5 and 20mm are completely removed using standard polypectomy snare. The investigation was also directed at a comparison between complete resection of polyps between 5 and 9mm and 10 and 20mm.

DETAILED DESCRIPTION:
All patients who present for a colonoscopy and meet inclusion and exclusion criteria will be asked to participate, and all patients with resectable polyps will be included. See also inclusion and exclusion criteria.

All patients will have undergone a regular bowel preparation with polyethylene glycol lavage with 4-6 L until clear rectal fluid is evacuated.

Polyp resection will be performed by experienced endoscopists (each with over 500 colonoscopies performed). All polyps between 5 and 20mm will be removed with an electro-cautery snare. Polyp size will be estimated using the snare catheter (2.5mm) or the snare diameter (10x20mm, 15x30mm, 20x20mm) before resection. The endoscopist will grade the difficulty of resection. Following the resection, the endoscopist will closely examine the resection margins. Biopsies will be taken from resection margins: 2 biopsies will be obtained from opposite margins for polyps 5-9mm, and 4 biopsies will be taken for polyps 10-20mm from all four quadrants of the resection margins. In case of assumed incomplete resection this will be documented and further (piecemeal) resections should be done, if this is not feasible, margins can be cauterized according to standard polypectomy resection (e.g. by argon beamer coagulation) after previous biopsy. Only those polyps that are found to be adenomatous polyps will be included in the analysis.

If polyp resection is complicated by bleeding (not self-sustained), no biopsies will be taken and any additional polyps that will be found during the remaining examination will be excluded from analysis. Any bleeding from the margins after polypectomy will be treated by endoscopic injection using diluted epinephrine (1:10.000).

A single research subject may have many eligible polyps. To avoid taking many biopsies, the investigators will not include more than 5 eligible polyps (the first 5 that are detected) per patient in the study.

Laboratory Analysis:

Polyps and biopsies will be sent to the pathology lab of each center. The polyps will be evaluated according to common practice. In addition information regarding resection margins will be provided for each polyp: R0= free of adenomatous tissue, R1=adenomatous tissue detected in the margin. This information is not routinely provided by the pathologist as there is so far no data whether this information is reliable. Only adenomatous polyps will be included in the analysis. Hyperplastic polyps will not be included. Biopsies will only be processed after the diagnosis of an adenomatous polyp was made. Biopsies will be evaluated for presence of adenomatous tissue. The additional impact for the pathology lab includes a) processing of biopsies belonging to the polyp specimens, and b) providing information on polyp margins. The VA pathology lab estimated the financial impact to be low and there will be no financial requests. The pathological diagnosis, including the reading of the biopsies, will become part of the medical record. If biopsies contain adenomatous tissue the patient will be ask to return for a follow-up colonoscopy within 1 year. This is within current standard of care to repeat a colonoscopy to assure complete adenoma resection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥40 and <85 who presents for a colonoscopy and does not meet any of the exclusion criteria mentioned below will be asked to participate
* All patients who are found to have colonic polyp between 5 and 20mm in size will be included in the study

Exclusion Criteria:

* Pedunculated polyps (estimated stalk diameter < 50% polyp head diameter, stalk at least 5 mm)
* Any suspicion of perforation or deeper defects after polypectomy, irrespective whether treated or not.
* Post-polypectomy bleeding requiring hemostasis.
* Patients with known inflammatory bowel disease or active colitis
* Patients who are receiving an emergency colonoscopy
* Poor general health (ASA class>3)
* Patients on coumadin or with coagulopathy with an elevated INR ≥1.8, or platelets <50.
* Poor bowel preparation
* Patients who do not consent
* Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants eligible for recruitment are patients who present for a colonoscopy to the VAMC or DHMC Gastroenterology department conducting this study. Upon arrival for a scheduled colonoscopy patient records will be reviewed to determine eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Pohl, MD, Principal Investigator — White River Junction VAMC, Dartmouth Medical School
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - White River Junction VAMC, White River Junction, Vermont

REFERENCES:
- [Derived] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1429 patients were consented, of which 269 met inclusion criteria.
Groups:
- All Adenomatous Polyps: Standard polypectomy snare of adenomatous polyps (included serrated adenomas) from ≥5mm to ≤20mm.
Period: Overall Study
Arm/Group | All Adenomatous Polyps
Started | 269
Completed | 269
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Adenomatous Polyps: Adenomatous polyps (included serrated adenomas) ≤5mm and ≤20mm.
Arm/Group | All Adenomatous Polyps
Number analyzed (Participants) | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 167
  >=65 years | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 226
Region of Enrollment [Number; unit: participants]
  United States | 269

OUTCOME MEASURES:

1. Primary Outcome: Percent of Incompletely Resected Adenomatous Polyps
Description: Proportion of incompletely resected adenomatous polyps (5 to 20mm), defined by remaining adenomatous tissue in marginal biopsies after snare resection.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of incomplete resection
Units Other Than Participants: N of adenomatous polyps
Groups:
- All Adenomatous Polyps: Adenomatous polyps (included serrated adenomas) ≥5mm and ≤20mm.
Arm/Group | All Adenomatous Polyps
Number analyzed (Participants) | 269
Number analyzed (N of adenomatous polyps) | 346
percentage of incomplete resection | 10.1 [6.9 to 13.3]

2. Secondary Outcome: Incomplete Adenoma Resection of Small and Large Adenomas
Description: Comparison of the proportion of incompletely resected adenomatous polyps by size (5-9mm versus 10-20mm).
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | All Adenomatous Polyps
Serious Adverse Events (participants affected / at risk) | 0/269
Other Adverse Events (participants affected / at risk) | 0/269

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No